CLINICAL TRIAL: NCT04657003
Title: Efficacy and Safety of Tirzepatide Once Weekly in Participants With Type 2 Diabetes Who Have Obesity or Are Overweight: A Randomized, Double-Blind, Placebo-Controlled Trial (SURMOUNT-2)
Brief Title: A Study of Tirzepatide (LY3298176) in Participants With Type 2 Diabetes Who Have Obesity or Are Overweight
Acronym: SURMOUNT-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17245; I8F-MC-GPHL (Other: Eli Lilly and Company)
Record Dates: First submitted 2020-12-01; First posted 2020-12-07 (Actual); Results first posted 2024-04-08 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-03

CONDITIONS: Type 2 Diabetes; Overweight; Obesity
Keywords: Metabolism and Nutrition Disorder
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Overweight; Obesity; Nutrition Disorders | interventions — Tirzepatide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 10 milligrams (mg) Tirzepatide (Experimental): 10 mg Tirzepatide administered subcutaneously (SC) once weekly (QW)
  Interventions: Drug: Tirzepatide
- 15 mg Tirzepatide (Experimental): 15 mg Tirzepatide administered SC QW
  Interventions: Drug: Tirzepatide
- Placebo (Placebo Comparator): Placebo administered SC QW
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Tirzepatide — Administered SC
  Other Names: LY3298176
  Arms: 10 milligrams (mg) Tirzepatide; 15 mg Tirzepatide
Other: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
This is a study of tirzepatide in participants with type 2 diabetes who have obesity or are overweight. The main purpose is to learn more about how tirzepatide affects body weight. The study will last 79 weeks (22 visits).

ELIGIBILITY:
Inclusion Criteria:

* Have Type 2 Diabetes (T2DM) with HbA1c ≥7% to ≤10% at screening, on stable therapy for the last 3 months prior to screening. T2DM may be treated with diet/exercise alone or any oral glycemic-lowering agent (as per local labeling) EXCEPT dipeptidyl peptidase 4 (DPP-4) inhibitors or glucagon like peptide-1 receptor agonists (GLP-1 RAs)
* Have a BMI of ≥27 kg/m²
* Are overweight or have obesity
* Have a history of at least 1 self-reported unsuccessful dietary effort to lose body weight
* Are at least 18 years of age and age of majority per local laws and regulations

Exclusion Criteria:

* Have Type 1 diabetes mellitus, history of ketoacidosis or hyperosmolar state/coma or any other types of diabetes except T2DM
* Have at least 2 confirmed fasting self-monitoring blood glucose (SMBG) values >270 mg/dL(on 2 nonconsecutive days) prior to Visit 3
* Have proliferative diabetic retinopathy OR diabetic macular edema OR non-proliferative diabetic retinopathy that requires acute treatment
* Have self-reported change in body weight >5kg within 3 months prior to screening
* Have had a history of chronic or acute pancreatitis
* Change in body weight greater than 5 kg within 3 months prior to starting study
* Obesity induced by other endocrinologic disorders or monogenetic or syndromic forms of obesity
* Family or personal history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia syndrome type 2 (MEN-2)
* History of significant active or unstable major depressive disorder (MDD) or other severe psychiatric disorder within the last 2 years
* Any lifetime history of a suicide attempt

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 938 (Actual)
Dates: Start 2021-03-29 (Actual); Primary Completion 2023-03-16 (Actual); Study Completion 2023-04-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (75):
- United States (43):
  - University of Alabama - Department of Nutrition Sciences, Birmingham, Alabama
  - KLR Business Group, Inc. dba Arkansas Clinical Research, Little Rock, Arkansas
  - Velocity Clinical Research, Huntington Park, Huntington Park, California
  - Velocity Clinical Research, Westlake, Los Angeles, California
  - Catalina Research Institute, LLC, Montclair, California
  - Encompass Clinical Research, Spring Valley, California
  - University Clinical Investigators, Inc., Tustin, California
  - ALL Medical Research, LLC, Cooper City, Florida
  - Northeast Research Institute (NERI), Fleming Island, Florida
  - New Horizon Research Center, Miami, Florida
  - West Orange Endocrinology, Ocoee, Florida
  - Metabolic Research Institute, Inc., West Palm Beach, Florida
  - Emory University School of Medicine- Grady Campus, Atlanta, Georgia
  - East Coast Institute for Research, LLC, Macon, Georgia
  - Pacific Diabetes & Endocrine Center, Honolulu, Hawaii
  - Elite Clinical Trials, Blackfoot, Idaho
  - Rocky Mountain Clinical Research, Idaho Falls, Idaho
  - American Health Network of Indiana, LLC - Greenfield, Greenfield, Indiana
  - Iowa Diabetes and Endocrinology Research Center, West Des Moines, Iowa
  - Cotton O'Neil Clinical Research Center, Topeka, Kansas
  - Maryland Cardiovascular Specialists, Baltimore, Maryland
  - MD Medical Research, Oxon Hill, Maryland
  - NECCR PrimaCare Research, Fall River, Massachusetts
  - Arcturus Healthcare , PLC, Troy Internal Medicine Research Division, Troy, Michigan
  - Logan Health Research, Kalispell, Montana
  - Premier Research, Trenton, New Jersey
  - University of North Carolina Medical Center, Chapel Hill, North Carolina
  - PharmQuest, Greensboro, North Carolina
  - Wake Forest University Baptist Medical Center (WFUBMC), Winston-Salem, North Carolina
  - Velocity Clinical Research, Cleveland, Cleveland, Ohio
  - Aventiv Research, Dublin, Ohio
  - The Corvallis Clinic, P.C., Corvallis, Oregon
  - Preferred Primary Care Physicians, Uniontown, Pennsylvania
  - Center for Neurosciences, Warwick, Rhode Island
  - Tribe Clinical Research, LLC, Greenville, South Carolina
  - Texas Diabetes & Endocrinology, P.A., Austin, Texas
  - Dallas Diabetes Research Center, Dallas, Texas
  - Diabetes and Thyroid Center of Fort Worth, Fort Worth, Texas
  - Juno Research, Houston, Texas
  - Endocrine Ips, Pllc, Houston, Texas
  - Health Research of Hampton Roads, Inc., Newport News, Virginia
  - Rainier Clinical Research Center, Renton, Washington
  - Clinical Investigation Specialists, Kenosha, Wisconsin
- Argentina (8):
  - Consultorio de Investigación Clínica EMO SRL, Ciudad Autonoma de Buenos Aire, Buenos Aires
  - Centro de Investigaciones Metabólicas (CINME), Ciudad Autónoma de Buenos Aire, Buenos Aires
  - Instituto de Investigaciones Clínicas Mar del Plata, Mar del Plata, Buenos Aires
  - Go Centro Medico San Nicolás, San Nicolás de los Arroyos, Buenos Aires
  - Centro Médico Viamonte, Buenos Aires, Ciudad Autónoma de Buenos Aire
  - CIPREC, CABA, Ciudad Autónoma de Buenos Aire
  - Centro de Investigaciones Médicas Tucuman, SAN M. de Tucuman, Tucumán Province
  - Sanatorio Norte, Santiago del Estero
- Brazil (6):
  - Private Practice - Dr.Miguel N. Hissa, Fortaleza, Ceará
  - Loema Instituto de Pesquisa Clinica, Campinas, São Paulo
  - Instituto de Pesquisa clinica de Campinas, Campinas, São Paulo
  - CECIP - Centro de Estudos do Interior Paulista, Jaú, São Paulo
  - CPCLIN, São Paulo, São Paulo
  - CEPIC - Centro Paulista de Investigação Clínica, São Paulo
- India (2):
  - Life Care Hospital and Research Centre, Bangalore, Karnataka
  - ILS Hospitals, Kolkata, West Bengal
- Japan (4):
  - Medical Corporation Yuga Tsuruma Kaneshiro Diabetes Clinic, Yamato-shi, Kanagawa
  - Medical Corporation Heishinkai OCROM Clinic, Suita-shi, Osaka
  - Medical Corporation Sato Medical clinic, Ootaku, Tokyo
  - AMC Nishiumeda Clinic, Osaka
- Puerto Rico (3):
  - Centro de Endocrinologia y Nutricion, Caguas
  - Latin Clinical Trial Center, San Juan
  - GCM Medical Group, PSC - Hato Rey Site, San Juan
- Russia (4):
  - Endocrinology Research Center of Rosmedtechnologies, Moscow, Moscow
  - Russian Medical Academy of Postgraduate Education, Moscow, Moscow
  - Saint-Petersburg City Hospital of Saint Elizabeth, Saint Petersburg, Sankt-Pete
  - Smolensk State Medical University, Smolensk
- Taiwan (5):
  - Changhua Christian Hospital, Changhua County, Changhua
  - Chi Mei Medical Center, Tainan, Tainan
  - Chung Shan Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Cheng-Kung Uni. Hosp., Tainan

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Time Frame:
  Data are available 6 months after the primary publication or approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://www.vivli.org/

REFERENCES:
- [Derived] Wadden TA, Oquendo MA, Kushner RF, Cao D, Karanikas CA, Kechter A, Murphy MA. Psychiatric Safety of Tirzepatide in People With Obesity and No Known Major Psychopathology: A Post Hoc Analysis of SURMOUNT. Obesity (Silver Spring). 2026 Jan 15. doi: 10.1002/oby.70122. Online ahead of print. PMID 41537305
- [Derived] Heerspink HJL, Friedman AN, Bjornstad P, van Raalte DH, Cherney D, Cao D, Garcia-Perez LE, Stefanski A, Turfanda I, Bunck MC, Benabbad I, Griffin R, Piras de Oliveira C. Kidney Parameters with Tirzepatide in Obesity with or without Type 2 Diabetes. J Am Soc Nephrol. 2025 Nov 1;36(11):2190-2200. doi: 10.1681/ASN.0000000764. Epub 2025 Jun 13. PMID 40512543
- [Derived] Hunter Gibble T, Cao D, Zhang XM, Xavier NA, Poon JL, Fitch A. Tirzepatide Was Associated with Improved Health-Related Quality of Life in Adults with Obesity or Overweight and Type 2 Diabetes: Results from the Phase 3 SURMOUNT-2 Trial. Diabetes Ther. 2025 May;16(5):977-991. doi: 10.1007/s13300-025-01723-w. Epub 2025 Mar 22. PMID 40120035
- [Derived] Garvey WT, Frias JP, Jastreboff AM, le Roux CW, Sattar N, Aizenberg D, Mao H, Zhang S, Ahmad NN, Bunck MC, Benabbad I, Zhang XM; SURMOUNT-2 investigators. Tirzepatide once weekly for the treatment of obesity in people with type 2 diabetes (SURMOUNT-2): a double-blind, randomised, multicentre, placebo-controlled, phase 3 trial. Lancet. 2023 Aug 19;402(10402):613-626. doi: 10.1016/S0140-6736(23)01200-X. Epub 2023 Jun 26. PMID 37385275
- See also: A Study of Tirzepatide (LY3298176) in Participants With Type 2 Diabetes Who Have Obesity or Are Overweight (SURMOUNT-2) — https://trials.lillytrialguide.com/en-US/trial/6Lso9L1WmsU8ly9DkEFiaU

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants received Placebo administered subcutaneously (SC) once weekly (QW).
- 10 Milligrams (mg) Tirzepatide: Participants received 10 mg Tirzepatide administered SC QW
- 15 mg Tirzepatide: Participants received 15 mg Tirzepatide administered SC QW
Period: Overall Study
Arm/Group | Placebo | 10 Milligrams (mg) Tirzepatide | 15 mg Tirzepatide
Started | 315 | 312 | 311
Received at Least One Dose of Study Drug | 315 | 312 | 311
Completed | 281 | 296 | 282
Not Completed | 34 | 16 | 29
Not completed — Adverse Event | 5 | 1 | 5
Not completed — Death | 0 | 2 | 0
Not completed — Lost to Follow-up | 8 | 4 | 10
Not completed — Other - As Reported by Investigator | 3 | 2 | 2
Not completed — Pregnancy | 2 | 0 | 2
Not completed — Withdrawal by Subject | 16 | 7 | 10

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Placebo: Participants received Placebo administered SC QW.
- 10 mg Tirzepatide: Participants received 10 mg Tirzepatide administered SC QW.
- Total: Total of all reporting groups
Arm/Group | Placebo | 10 mg Tirzepatide | 15 mg Tirzepatide | Total
Number analyzed (Participants) | 315 | 312 | 311 | 938
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.7 (10.5) | 54.3 (10.7) | 53.6 (10.6) | 54.2 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 159 | 158 | 159 | 476
  Male | 156 | 154 | 152 | 462
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 188 | 184 | 189 | 561
  Not Hispanic or Latino | 122 | 124 | 112 | 358
  Unknown or Not Reported | 5 | 4 | 10 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 39 | 44 | 42 | 125
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 1 | 3
  Black or African American | 22 | 33 | 22 | 77
  White | 248 | 228 | 234 | 710
  More than one race | 5 | 6 | 12 | 23
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Argentina | 116 | 115 | 115 | 346
  Brazil | 30 | 29 | 30 | 89
  India | 9 | 8 | 9 | 26
  Japan | 21 | 24 | 22 | 67
  Russia | 17 | 13 | 13 | 43
  Taiwan | 8 | 9 | 8 | 25
  United States | 114 | 114 | 114 | 342
Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 101.65 (22.26) | 100.86 (20.93) | 99.60 (20.05) | 100.71 (21.10)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Body Weight
Description: Least Squares Mean (LSMean) calculated using Mixed Model Repeated Measures (MMRM) model for post-baseline measures: Variable = Baseline + Analysis Country + Sex + Type of Antihyperglycemic Medication (AHM) Used at Randomization + Treatment + Time + Treatment*Time (Type III sum of squares).
Time Frame: Baseline, Week 72
Population: All randomized participants who received at least one dose of study drug. Only participants with non-missing baseline value and at least one non-missing post-baseline value of the response variable were included in analysis.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | 10 mg Tirzepatide | 15 mg Tirzepatide
Number analyzed (Participants) | 311 | 309 | 309
percent change | -3.3 (0.49) | -13.4 (0.48) | -15.7 (0.49)
Statistical Analysis 1: Comparison: Placebo vs 10 mg Tirzepatide; Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Mean Difference (Net) = -10.1, 95% CI 2-sided [-11.5 to -8.8]
Statistical Analysis 2: Comparison: Placebo vs 15 mg Tirzepatide; Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Mean Difference (Net) = -12.4, 95% CI 2-sided [-13.7 to -11.0]

2. Primary Outcome: Percentage of Participants Who Achieve ≥5% Body Weight Reduction From Baseline
Description: Percentage of participants who achieve ≥5% body weight reduction from baseline
Time Frame: Week 72
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 10 mg Tirzepatide | 15 mg Tirzepatide
Number analyzed (Participants) | 311 | 309 | 309
percentage of participants | 30.55 | 81.55 | 86.41
Statistical Analysis 1: Comparison: Placebo vs 10 mg Tirzepatide; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 10.75, 95% CI 2-sided [7.30 to 15.84]
Statistical Analysis 2: Comparison: Placebo vs 15 mg Tirzepatide; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 15.28, 95% CI 2-sided [10.08 to 23.14]

3. Secondary Outcome: Percentage of Participants Who Achieve ≥10% Body Weight Reduction From Baseline
Description: Percentage of participants who achieve ≥10% body weight reduction from baseline
Time Frame: Week 72
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 10 mg Tirzepatide | 15 mg Tirzepatide
Number analyzed (Participants) | 311 | 309 | 309
percentage of participants | 8.68 | 63.43 | 69.58
Statistical Analysis 1: Comparison: Placebo vs 10 mg Tirzepatide; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 20.94, 95% CI 2-sided [13.06 to 33.58]
Statistical Analysis 2: Comparison: Placebo vs 15 mg Tirzepatide; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 27.50, 95% CI 2-sided [17.04 to 44.39]

4. Secondary Outcome: Percentage of Participants Who Achieve ≥15% Body Weight Reduction From Baseline
Description: Percentage of participants who achieve ≥15% body weight reduction from baseline
Time Frame: Week 72
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 10 mg Tirzepatide | 15 mg Tirzepatide
Number analyzed (Participants) | 311 | 309 | 309
percentage of participants | 2.57 | 41.42 | 51.78
Statistical Analysis 1: Comparison: Placebo vs 10 mg Tirzepatide; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 28.38, 95% CI 2-sided [13.81 to 58.31]
Statistical Analysis 2: Comparison: Placebo vs 15 mg Tirzepatide; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 43.60, 95% CI 2-sided [21.20 to 89.67]

5. Secondary Outcome: Percentage of Participants Who Achieve ≥20% Body Weight Reduction From Baseline
Description: Percentage of participants who achieve ≥20% body weight reduction from baseline
Time Frame: Week 72
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 10 mg Tirzepatide | 15 mg Tirzepatide
Number analyzed (Participants) | 311 | 309 | 309
percentage of participants | 0.96 | 22.98 | 33.98
Statistical Analysis 1: Comparison: Placebo vs 10 mg Tirzepatide; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 28.54, 95% CI 2-sided [9.73 to 83.73]
Statistical Analysis 2: Comparison: Placebo vs 15 mg Tirzepatide; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 49.68, 95% CI 2-sided [17.03 to 144.94]

6. Secondary Outcome: Change From Baseline in Absolute Body Weight
Description: LSMean calculated using MMRM model for post-baseline measures: Variable = Baseline + Analysis Country + Sex + Type of AHM Used at Randomization + Treatment + Time + Treatment*Time (Type III sum of squares).
Time Frame: Baseline, Week 72
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: kilograms (kg)
Arm/Group | Placebo | 10 mg Tirzepatide | 15 mg Tirzepatide
Number analyzed (Participants) | 311 | 309 | 309
kilograms (kg) | -3.2 (0.51) | -13.5 (0.51) | -15.6 (0.51)
Statistical Analysis 1: Comparison: Placebo vs 10 mg Tirzepatide; Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Mean Difference (Net) = -10.3, 95% CI 2-sided [-11.7 to -8.8]
Statistical Analysis 2: Comparison: Placebo vs 15 mg Tirzepatide; Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Mean Difference (Net) = -12.4, 95% CI 2-sided [-13.8 to -11.0]

7. Secondary Outcome: Change From Baseline in Body Mass Index (BMI)
Description: as for outcome 6
Time Frame: Baseline, Week 72
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: kilograms per meter squared (kg/m^2)
Arm/Group | Placebo | 10 mg Tirzepatide | 15 mg Tirzepatide
Number analyzed (Participants) | 311 | 309 | 309
kilograms per meter squared (kg/m^2) | -1.2 (0.19) | -4.9 (0.18) | -5.7 (0.19)
Statistical Analysis 1: Comparison: Placebo vs 10 mg Tirzepatide; Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Mean Difference (Net) = -3.7, 95% CI 2-sided [-4.2 to -3.2]
Statistical Analysis 2: Comparison: Placebo vs 15 mg Tirzepatide; Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Mean Difference (Net) = -4.5, 95% CI 2-sided [-5.0 to -4.0]

8. Secondary Outcome: Change From Baseline in Hemoglobin A1c (HbA1c)
Description: as for outcome 6
Time Frame: Baseline, Week 72
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | Placebo | 10 mg Tirzepatide | 15 mg Tirzepatide
Number analyzed (Participants) | 290 | 301 | 300
percentage of HbA1c | -0.16 (0.067) | -2.14 (0.060) | -2.22 (0.060)
Statistical Analysis 1: Comparison: Placebo vs 10 mg Tirzepatide; Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Mean Difference (Net) = -1.97, 95% CI 2-sided [-2.15 to -1.80]
Statistical Analysis 2: Comparison: Placebo vs 15 mg Tirzepatide; Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Mean Difference (Net) = -2.06, 95% CI 2-sided [-2.24 to -1.88]

9. Secondary Outcome: Percentage of Participants Who Achieve HbA1c <7%
Description: Percentage of participants who achieve HbA1c <7%
Time Frame: Week 72
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 10 mg Tirzepatide | 15 mg Tirzepatide
Number analyzed (Participants) | 290 | 301 | 300
percentage of participants | 29.31 | 90.03 | 90.67
Statistical Analysis 1: Comparison: Placebo vs 10 mg Tirzepatide; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 28.01, 95% CI 2-sided [17.21 to 45.59]
Statistical Analysis 2: Comparison: Placebo vs 15 mg Tirzepatide; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 34.19, 95% CI 2-sided [20.27 to 57.67]

10. Secondary Outcome: Percentage of Participants Who Achieve HbA1c ≤6.5%
Description: Percentage of participants who achieve HbA1c ≤6.5%
Time Frame: Week 72
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 10 mg Tirzepatide | 15 mg Tirzepatide
Number analyzed (Participants) | 290 | 301 | 300
percentage of participants | 15.52 | 84.05 | 86.67
Statistical Analysis 1: Comparison: Placebo vs 10 mg Tirzepatide; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 42.11, 95% CI 2-sided [25.61 to 69.26]
Statistical Analysis 2: Comparison: Placebo vs 15 mg Tirzepatide; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 58.67, 95% CI 2-sided [34.29 to 100.37]

11. Secondary Outcome: Percentage of Participants Who Achieve HbA1c <5.7%
Description: Percentage of participants who achieve HbA1c <5.7%
Time Frame: Week 72
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | 10 mg Tirzepatide | 15 mg Tirzepatide
Number analyzed (Participants) | 290 | 301 | 300
percentage of participants | 2.76 | 50.17 | 55.33
Statistical Analysis 1: Comparison: Placebo vs 10 mg Tirzepatide; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 42.55, 95% CI 2-sided [20.46 to 88.50]
Statistical Analysis 2: Comparison: Placebo vs 15 mg Tirzepatide; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 54.30, 95% CI 2-sided [26.00 to 113.38]

12. Secondary Outcome: Change From Baseline in Fasting Glucose
Description: LSMean calculated using MMRM model for post-baseline measures: Variable = Baseline + Analysis Country + Sex + Type of AHM Used at Randomization + Baseline HbA1c Group (<=8.5%, >8.5%) + Treatment + Time + Treatment*Time (Type III sum of squares).
Time Frame: Baseline, Week 72
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: milligrams per deciliter (mg/dL)
Arm/Group | Placebo | 10 mg Tirzepatide | 15 mg Tirzepatide
Number analyzed (Participants) | 290 | 300 | 300
milligrams per deciliter (mg/dL) | -2.42 (2.281) | -49.20 (1.940) | -51.67 (1.970)
Statistical Analysis 1: Comparison: Placebo vs 10 mg Tirzepatide; Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Mean Difference (Net) = -46.79, 95% CI 2-sided [-52.67 to -40.91]
Statistical Analysis 2: Comparison: Placebo vs 15 mg Tirzepatide; Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Mean Difference (Net) = -49.25, 95% CI 2-sided [-55.18 to -43.33]

13. Secondary Outcome: Change From Baseline in Waist Circumference
Description: as for outcome 6
Time Frame: Baseline, Week 72
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: centimeters (cm)
Arm/Group | Placebo | 10 mg Tirzepatide | 15 mg Tirzepatide
Number analyzed (Participants) | 311 | 309 | 309
centimeters (cm) | -3.4 (0.51) | -11.2 (0.50) | -13.8 (0.51)
Statistical Analysis 1: Comparison: Placebo vs 10 mg Tirzepatide; Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Mean Difference (Net) = -7.8, 95% CI 2-sided [-9.2 to -6.4]
Statistical Analysis 2: Comparison: Placebo vs 15 mg Tirzepatide; Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Mean Difference (Net) = -10.4, 95% CI 2-sided [-11.8 to -8.9]

14. Secondary Outcome: Percent Change From Baseline in Total Cholesterol (Pooled Doses of Tirzepatide 10 mg and 15 mg)
Description: Results are reported as model-based estimates and standard error (SE) from MMRM analysis using log transformation.
Time Frame: Baseline, Week 72
Population: All randomized participants who received at least one dose of study drug. Only participants with non-missing baseline value and at least one non-missing post-baseline value of the response variable were included in analysis. This analysis was planned to measure the outcome data under a single arm (pooled 10 mg and 15 mg Tirzepatide).
Measure: Mean (Standard Error); unit: percent change
Groups:
- Pooled 10 mg and 15 mg Tirzepatide: Participants received Tirzepatide administered SC QW. Participants in 10 mg and 15 mg Tirzepatide arms were pooled in this arm.
Arm/Group | Placebo | Pooled 10 mg and 15 mg Tirzepatide
Number analyzed (Participants) | 292 | 587
percent change | 2.13 (1.135) | -2.58 (0.755)
Statistical Analysis 1: Comparison: Placebo vs Pooled 10 mg and 15 mg Tirzepatide; Test type: Superiority; p < 0.001, Mixed Models Analysis; Estimate Difference = -4.61, 95% CI 2-sided [-7.11 to -2.03]

15. Secondary Outcome: Percent Change From Baseline in Low Density Lipoprotein (LDL) Cholesterol (Pooled Doses of Tirzepatide 10 mg and 15 mg)
Description: Results are reported as model-based estimates and SE from MMRM analysis using log transformation.
Time Frame: Baseline, Week 72
Population: as for outcome 14
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Pooled 10 mg and 15 mg Tirzepatide
Number analyzed (Participants) | 292 | 587
percent change | 6.29 (1.874) | 2.72 (1.264)
Statistical Analysis 1: Comparison: Placebo vs Pooled 10 mg and 15 mg Tirzepatide; Test type: Superiority; p = 0.112, Mixed Models Analysis; Estimate Difference = -3.36, 95% CI 2-sided [-7.36 to 0.81]

16. Secondary Outcome: Percent Change From Baseline in High Density Lipoprotein (HDL) Cholesterol (Pooled Doses of Tirzepatide 10 mg and 15 mg)
Description: Results are reported as model-based estimates and SE from MMRM analysis using log transformation.
Time Frame: Baseline, Week 72
Population: as for outcome 14
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Pooled 10 mg and 15 mg Tirzepatide
Number analyzed (Participants) | 292 | 587
percent change | 1.10 (1.048) | 8.19 (0.782)
Statistical Analysis 1: Comparison: Placebo vs Pooled 10 mg and 15 mg Tirzepatide; Test type: Superiority; p < 0.001, Mixed Models Analysis; Estimate Difference = 7.02, 95% CI 2-sided [4.40 to 9.71]

17. Secondary Outcome: Percent Change From Baseline in Very Low Density Lipoprotein (VLDL) Cholesterol (Pooled Doses of Tirzepatide 10 mg and 15 mg)
Description: Results are reported as model-based estimates and SE from MMRM analysis using log transformation.
Time Frame: Baseline, Week 72
Population: as for outcome 14
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Pooled 10 mg and 15 mg Tirzepatide
Number analyzed (Participants) | 284 | 574
percent change | -6.0 (2.18) | -27.9 (1.16)
Statistical Analysis 1: Comparison: Placebo vs Pooled 10 mg and 15 mg Tirzepatide; Test type: Superiority; p < 0.001, Mixed Models Analysis; Estimate Difference = -23.3, 95% CI 2-sided [-27.5 to -18.9]

18. Secondary Outcome: Percent Change From Baseline in Triglycerides (Pooled Doses of Tirzepatide 10 mg and 15 mg)
Description: Results are reported as model-based estimates and SE from MMRM analysis using log transformation.
Time Frame: Baseline, Week 72
Population: as for outcome 14
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Pooled 10 mg and 15 mg Tirzepatide
Number analyzed (Participants) | 292 | 587
percent change | -5.8 (2.32) | -28.6 (1.22)
Statistical Analysis 1: Comparison: Placebo vs Pooled 10 mg and 15 mg Tirzepatide; Test type: Superiority; p < 0.001, Mixed Models Analysis; Estimate Difference = -24.2, 95% CI 2-sided [-28.6 to -19.6]

19. Secondary Outcome: Percent Change From Baseline in Non-High Density Lipoprotein (Non-HDL) Cholesterol (Pooled Doses of Tirzepatide 10 mg and 15 mg)
Description: Results are reported as model-based estimates and SE from MMRM analysis using log transformation.
Time Frame: Baseline, Week 72
Population: as for outcome 14
Measure: Mean (Standard Error); unit: percent change
Groups:
- Pooled Doses of 10 mg and 15 mg Tirzepatide: Participants received Tirzepatide administered SC QW. Participants in 10 mg and 15 mg Tirzepatide arms were pooled in this arm.
Arm/Group | Placebo | Pooled Doses of 10 mg and 15 mg Tirzepatide
Number analyzed (Participants) | 292 | 587
percent change | 2.30 (1.573) | -6.64 (1.001)
Statistical Analysis 1: Comparison: Placebo vs Pooled Doses of 10 mg and 15 mg Tirzepatide; Test type: Superiority; p < 0.001, Mixed Models Analysis; Estimate Difference = -8.74, 95% CI 2-sided [-12.04 to -5.32]

20. Secondary Outcome: Percent Change From Baseline in Free Fatty Acids (Pooled Doses of 10 mg and 15 mg Tirzepatide)
Description: Results are reported as model-based estimates and SE from MMRM analysis using log transformation.
Time Frame: Baseline, Week 72
Population: as for outcome 14
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Pooled 10 mg and 15 mg Tirzepatide
Number analyzed (Participants) | 291 | 586
percent change | 0.03 (2.838) | -23.58 (1.502)
Statistical Analysis 1: Comparison: Placebo vs Pooled 10 mg and 15 mg Tirzepatide; Test type: Superiority; p < 0.001, Mixed Models Analysis; Estimate Difference = -23.61, 95% CI 2-sided [-28.62 to -18.24]

21. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) (Pooled Doses of 10 mg and 15 mg Tirzepatide)
Description: LSMean was calculated using MMRM model for post-baseline measures: Variable = Baseline + Analysis Country + Sex + Type of AHM Used at Randomization + Treatment + Time + Treatment*Time (Type III sum of squares).
Time Frame: Baseline, Week 72
Population: as for outcome 14
Measure: Least Squares Mean (Standard Error); unit: millimeters of mercury (mmHg)
Arm/Group | Placebo | Pooled 10 mg and 15 mg Tirzepatide
Number analyzed (Participants) | 311 | 618
millimeters of mercury (mmHg) | -1.0 (0.74) | -7.2 (0.52)
Statistical Analysis 1: Comparison: Placebo vs Pooled 10 mg and 15 mg Tirzepatide; Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Mean Difference (Net) = -6.2, 95% CI 2-sided [-8.0 to -4.4]

22. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure (DBP) (Pooled Doses of 10 mg and 15 mg Tirzepatide)
Description: as for outcome 21
Time Frame: Baseline, Week 72
Population: as for outcome 14
Measure: Least Squares Mean (Standard Error); unit: millimeters of mercury (mmHg)
Arm/Group | Placebo | Pooled Doses of 10 mg and 15 mg Tirzepatide
Number analyzed (Participants) | 311 | 618
millimeters of mercury (mmHg) | -0.2 (0.45) | -2.6 (0.31)
Statistical Analysis 1: Comparison: Placebo vs Pooled Doses of 10 mg and 15 mg Tirzepatide; Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Mean Difference (Net) = -2.4, 95% CI 2-sided [-3.5 to -1.3]

23. Secondary Outcome: Percent Change From Baseline in Fasting Insulin
Description: Results are reported as model-based estimates and SE from MMRM analysis using log transformation.
Time Frame: Baseline, Week 72
Population: as for outcome 1
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Placebo | 10 mg Tirzepatide | 15 mg Tirzepatide
Number analyzed (Participants) | 247 | 282 | 280
percent change | -14.5 (3.39) | -29.6 (2.28) | -40.3 (1.99)
Statistical Analysis 1: Comparison: Placebo vs 10 mg Tirzepatide; Test type: Superiority; p < 0.001, Mixed Models Analysis; Estimate Difference = -17.6, 95% CI 2-sided [-25.5 to -8.9]
Statistical Analysis 2: Comparison: Placebo vs 15 mg Tirzepatide; Test type: Superiority; p < 0.001, Mixed Models Analysis; Estimate Difference = -30.2, 95% CI 2-sided [-37.0 to -22.7]

24. Secondary Outcome: Change From Baseline in Short Form 36 Health Survey Version 2 (SF-36v2) Acute Form Physical Functioning Domain Score
Description: The SF-36v2 acute, 1-week recall version is a 36-item, generic, patient-administered measure designed to assess the following 8 domains: Physical Functioning, Role-Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role-Emotional, and Mental Health. The Physical-Functioning domain assesses limitations due to health "now" while the remaining domains assess functioning "in the past week." Each domain is scored individually and information from these 8 domains are further aggregated into 2 health-component summary scores: Physical-Component Summary and Mental-Component Summary. Items are answered on Likert scales of varying lengths (3-, 5-, or 6- point scales).The summary scores range from 0 to 100, with higher scores indicating better levels of function and/or better health.
Time Frame: Baseline, Week 72
Population: All randomized participants who received at least one dose of study drug. Only participants with non-missing baseline value and at least one non-missing post-baseline value of the response variable were included in analysis. Missing data was imputed using Last Observation Carried Forward (LOCF) method.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | 10 mg Tirzepatide | 15 mg Tirzepatide
Number analyzed (Participants) | 270 | 281 | 270
score on a scale | 1.6 (0.40) | 3.4 (0.39) | 3.8 (0.40)
Statistical Analysis 1: Comparison: Placebo vs 10 mg Tirzepatide; Test type: Superiority; p = 0.001, ANCOVA; LSMean Mean Difference (Net) = 1.8, 95% CI 2-sided [0.7 to 2.9]
Statistical Analysis 2: Comparison: Placebo vs 15 mg Tirzepatide; Test type: Superiority; p < 0.001, ANCOVA; LSMean Mean Difference (Net) = 2.3, 95% CI 2-sided [1.1 to 3.4]

25. Secondary Outcome: Change From Baseline in Impact of Weight on Quality of Life-Lite-Clinical Trials Version (IWQOL Lite-CT) Physical Function Composite Score
Description: The IWQOL-Lite-CT is a 20-item, obesity-specific patient reported outcome (PRO) instrument developed for use in obesity clinical trials. It assesses 2 primary domains of obesity-related health-related quality of life (HRQoL): physical (7 items), and psychosocial (13 items). A 5-item subset of the physical domain, the physical-function composite is also supported. Items in the physical-function composite describe physical impacts related to general and specific physical activities. All items in the physical domain are rated on either a 5-point frequency ("never" to "always") scale or a 5-point truth ("not at all true" to "completely true") scale. Total score of IWQOL-Lite-CT composite ranges from 0 to 100, with higher scores reflecting better quality of life.
Time Frame: Baseline, Week 72
Population: as for outcome 24
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | 10 mg Tirzepatide | 15 mg Tirzepatide
Number analyzed (Participants) | 270 | 282 | 269
score on a scale | 7.4 (1.03) | 14.3 (1.00) | 15.2 (1.03)
Statistical Analysis 1: Comparison: Placebo vs 10 mg Tirzepatide; Test type: Superiority; p < 0.001, ANCOVA; LSMean Difference (Net) = 6.9, 95% CI 2-sided [4.1 to 9.7]
Statistical Analysis 2: Comparison: Placebo vs 15 mg Tirzepatide; Test type: Superiority; p < 0.001, ANCOVA; LSMean Difference (Net) = 7.8, 95% CI 2-sided [5.0 to 10.7]

26. Secondary Outcome: Population Pharmacokinetics (PopPK): Steady State Area Under the Concentration Curve (AUC) of Tirzepatide
Description: Each participant was assigned via the Interactive Web Response System (IWRS) to one of the sampling PK time windows of 1 to 24 hours, 24 to 96 hours, or 120 to 168 hours postdose. The steady state AUC was evaluated using Population PK modeling.
Time Frame: Week 8, 16, 36: 1 to 24 hours, 24 to 96 hours, or 120 to 168 hours postdose
Population: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour per milliliter (ng*h/mL)
Arm/Group | 10 mg Tirzepatide | 15 mg Tirzepatide
Number analyzed (Participants) | 308 | 308
nanograms*hour per milliliter (ng*h/mL) | 153000 (19.5) | 234000 (19.2)

ADVERSE EVENTS:
Time Frame: Baseline through Week 76
Description: All participants who received at least one dose of study drug. Gender specific events only occurring in male or female participants have had the number of participants At Risk adjusted accordingly.
Arm/Group | Placebo | 10 mg Tirzepatide | 15 mg Tirzepatide
All-Cause Mortality (participants affected / at risk) | 0/315 | 2/312 | 0/311
Serious Adverse Events (participants affected / at risk) | 23/315 | 18/312 | 27/311
Other Adverse Events (participants affected / at risk) | 158/315 | 169/312 | 159/311
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo (N=315) | 10 mg Tirzepatide (N=312) | 15 mg Tirzepatide (N=311)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (3) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hernial eventration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Inguinal hernia strangulated (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Obstructive pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 2 (2) | 1 (1) | 2 (2)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 2 (2)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Appendicitis perforated (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Covid-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Covid-19 pneumonia (Infections and infestations) | 2 (3) | 0 (0) | 1 (1)
Gangrene (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Limb traumatic amputation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Post procedural haematuria (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Respiratory fume inhalation disorder (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Shunt thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/159 (0) | 0/158 (0) | 1/159 (1)
Gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Mantle cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/156 (0) | 0/154 (0) | 1/152 (1)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 3 (3) | 0 (0)
Calculus bladder (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Adenomyosis (Reproductive system and breast disorders) | 0/159 (0) | 1/158 (1) | 0/159 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral venous disease (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=315) | 10 mg Tirzepatide (N=312) | 15 mg Tirzepatide (N=311)
Abdominal pain (Gastrointestinal disorders) | 7 (17) | 12 (16) | 23 (31)
Constipation (Gastrointestinal disorders) | 13 (16) | 25 (31) | 28 (40)
Diarrhoea (Gastrointestinal disorders) | 28 (40) | 62 (127) | 66 (180)
Dyspepsia (Gastrointestinal disorders) | 10 (14) | 23 (30) | 22 (50)
Eructation (Gastrointestinal disorders) | 2 (3) | 19 (31) | 13 (23)
Nausea (Gastrointestinal disorders) | 20 (23) | 63 (250) | 68 (157)
Vomiting (Gastrointestinal disorders) | 10 (13) | 34 (56) | 40 (60)
Covid-19 (Infections and infestations) | 53 (55) | 52 (55) | 33 (33)
Nasopharyngitis (Infections and infestations) | 17 (22) | 9 (10) | 10 (12)
Upper respiratory tract infection (Infections and infestations) | 21 (28) | 10 (16) | 12 (14)
Decreased appetite (Metabolism and nutrition disorders) | 7 (7) | 30 (32) | 31 (40)
Hyperglycaemia (Metabolism and nutrition disorders) | 45 (46) | 6 (6) | 4 (4)
Dizziness (Nervous system disorders) | 5 (5) | 17 (19) | 8 (10)
Headache (Nervous system disorders) | 9 (14) | 16 (27) | 15 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-11-23): https://cdn.clinicaltrials.gov/large-docs/03/NCT04657003/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-13): https://cdn.clinicaltrials.gov/large-docs/03/NCT04657003/SAP_001.pdf